CLINICAL TRIAL: NCT03412279
Title: Translation, Cross-cultural Adaptation, and Psychometric Properties of the Hausa Versions of the Oswestry Disability Index, Numeric Pain Rating Scale, Roland-Morris Disability Questionnaire, SF-12 Health Survey, Pain Catastrophizing Scale, Fear-Avoidance Beliefs Questionnaire, Global Rating of Change Scale and Back Beliefs Questionnaire in Patients With Low Back Pain
Brief Title: Validation of Hausa Oswestry Disability Index, Numeric Pain Rating Scale, Roland-Morris Disability Questionnaire, SF-12 Health Survey, Pain Catastrophizing Scale, Fear-Avoidance Beliefs Questionnaire,Global Rating of Change Scale and Back Beliefs Questionnaire in Low Back Pain Patients
Status: Completed | Type: Observational
Sponsor: Bayero University Kano, Nigeria (Other)
Responsible Party: Principal Investigator, Aminu A. Ibrahim, Principal Investigator, Bayero University Kano, Nigeria
Other Study IDs: PPT/00009
Record Dates: First submitted 2018-01-15; First posted 2018-01-26 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Chronic Low Back Pain
Keywords: Chronic Low Back Pain; Oswestry Disability Index; Numeric Pain Rating Scale; Roland Morris Disability Questionnaire; SF-12 Health Survey; Fear-Avoidance Beliefs Questionnaire; Pain Catastrophizing Scale; Global Rating of Change Scale; Back Beliefs Questionnaire

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Application of the initial evaluation — Initial evaluation involves the application of Hausa ODI, NPRS, RMDQ, SF-12, PCS, GROC, BBQ, VAS for pain and disability, and FFD.
Behavioral: Final application of instruments — Application of the Hausa versions of ODI, NPRS, RMDQ, SF-12, PCS, GROC and BBQ one week after initial evaluation

SUMMARY:
Oswestry Disability Index (ODI), Numeric Pain Rating Scale, Roland-Morris Disability Questionnaire (RMDQ), SF-12 Health Survey, Pain Catastrophizing Scale (PCS), Fear-Avoidance Beliefs Questionnaire (FABQ), Global Rating of Change Scale and Back Beliefs Questionnaire (BBQ) are important and widely used validated patient self-reported measures commonly used in clinical trials and health research involving patients with low back pain (LBP). However, to date, validated Hausa versions of these tools are unavailable for use despite not only Hausa language is commonly spoken in Nigeria but in other parts of the world.

The purpose of this study is to perform, using evidence-based guidelines, translation, cultural adaptation and validation of the ODI, NPRS, RMDQ, SF-12 health survey, FABQ, PCS, GROC and BBQ into Hausa language among patients with LBP in Northern Nigeria.

DETAILED DESCRIPTION:
This study will test the psychometric properties (i.e validity; reliability, and ceiling effect) of the ODI-H, NPRS, RMDQ-H, SF-12-H, FABQ-H, PCS-H, GROC and BBQ-H in Hausa-speaking patients with LBP. Rural and urban participants with LBP will be recruited purposively. Copies of the translated Hausa versions of the NPRS, ODI, RMDQ, SF-12, FABQ, PCS, BBQ as well as VAS for pain and disability will be self or interviewer-administered. Lumbopelvic mobility using finger-floor distance test (FFD) will be also measured. The Hausa versions of the ODI, NPRS, RMDQ, SF-12, FABQ, PCS, GROC and BBQ will be administered again a week after.

Data will be analysed using descriptive, correlation, and factorial analysis on IBM SPSS (version 23.0) at alpha level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Male and female between 18 and 70 years old.
* Nonspecific low back pain lasting for more than 12 weeks.
* Resident in the selected rural and urban communities in Kano State Nigeria.
* Ability to read/understand English or Hausa language.

Exclusion Criteria:

* Previous history of back surgery.
* Spine pathology (e.g. tumor, infection, fracture)
* Severe cognitive impairment
* Impaired capacity to be interviewed
* Current pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with CLBP attending either rural or urban physiotherapy clinics in Kano State, Northern Nigeria.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Change in functional disability | Baseline and 1 week after baseline
  Functional disability will be measured by the Hausa Oswestry disability index (ODI-H). The questionnaire consists of 10 items with each item having six statements. All scores are summed, then multiplied by two to obtain the index (range 0 to 100) with higher score indicating greater disability.
Change in pain intensity | Baseline and 1 week after baseline
  Pain intensity will be measured by the Hausa Numeric Pain Rating Scale (NPRS-H). The score ranges from 0 to 10, with 0 indicating "No Pain" and 10 "Worst Imaginable Pain".
Change in functional disability | Baseline and 1 week after baseline
  Functional disability will be measured by the Hausa Roland-Morris Disability Questionnaire (RMDQ-H). The score ranges from 0 to 24, with 0 indicating no disability and 24 maximum disability.
Change in quality of life | Baseline and 1 week after baseline
  Quality of life will be measured using the Hausa SF-12 Health Hurvey (SF-12-H). The questionnaire consists of 12 items questioned weighted and summed to provide physical and mental health scores (PCS and MCS). The two composite scores are computed using the scores on twelve questions that range from 0 to 100, with higher score indicating better health.
Change in fear-avoidance beliefs | Baseline and 1 week after baseline
  Fear-avoidance beliefs will be measured by the Hausa fear avoidance beliefs
Change in pain catastrophization | Baseline and 1 week after baseline
  Pain catastrophization will be measured by the Hausa Pain Catastrophizing Scale (PCS-H). The scale consists of 13 items rated on 5-point ordinal scale (0-5).The total score ranges from 0-52 with higher score indicating more catastrophic thoughts.
Change in back beliefs | Baseline and 1 week after baseline
  Back pain beliefs will be evaluated by the Hausa Back Beliefs Questionnaire (BBQ-H). The questionnaire consists of 14 items with 9 items ranked on a 5 point scale and used to calculate a final score from 9 to 45. Higher scores are indicative of better LBP beliefs and indicate the potential of a better ability to cope with LBP.
Change in perceived recovery | Baseline and 1 week after baseline
  Perceived recovery will be evaluated by the Hausa Global Rating Change of Scale (GROC-H). The scale is an 11-point scale ranging from -5 to +5 with a mid-point (0) representing " no change", a left anchor (-5) representing "Very much Worse" and a right anchor (+5) representing "Completely Recovered".

SECONDARY OUTCOMES:
Change in pain Intensity | Baseline only
  Pain Intensity will be measured by 100 mm Visual Analogue Scale (VAS-P), in which 0 represents "no pain" and 10 represents "worst pain imaginable".
Change in disability | Baseline only
  Disability will be measured by 100 mm Visual Analogue Scale (VAS-D), in which 0 represents "no disability" and 10 represents "severe disability".
Change in mobility of the spine and pelvis | Baseline only
  The finger-floor distance test (FFD) measures mobility of both the whole spine and the pelvis in the overall motion of bending forward.

CONTACTS AND LOCATIONS:
Locations (1):
- Murtala Muhammad Specialist Hospital, Wudil General Hospital, Rano General Hospital, Kura General Hospital, and Dawakin-Kudu General Hospital, Kano, Nigeria

IPD SHARING:
Plan to Share IPD: Undecided